CLINICAL TRIAL: NCT03851666
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Exploratory Study to Assess the Effect of a Once Daily Administration of a Plant-based Hydrolysates in the Reduction of Hb1A) Levels in Pre-diabetic Volunteers.
Brief Title: Effect of a Plant-based Hydrolysates Daily Consumption on the HbA1c of Pre-diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onorach Clinical Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRT-pep-DB-01
Record Dates: First submitted 2019-02-15; First posted 2019-02-22 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12 weeks daily administration Placebo (Placebo Comparator): Intervention: 12 weeks daily administration. The placebo is a powder: microcrystalline cellulose. The daily dose administrated is 15 grams.
  Interventions: Other: 12 weeks daily administration Placebo
- 12 weeks daily administration Cereal 1 (Experimental): Intervention: 12 weeks daily administration. The plant-based hydrolysate is a powder. The product results from an extraction of the protein of a cereal (Cereal 1).
  The daily dose administrated is 15 grams.
  Interventions: Dietary Supplement: 12 weeks daily administration Cereal 1
- 12 weeks daily administration Cereal 2 (Active Comparator): Intervention: 12 weeks daily administration. The plant-based hydrolysate is a powder. The product results from an extraction of the protein of a cereal (Cereal 2).
  The daily dose administrated is 15 grams.
  Interventions: Dietary Supplement: 12 weeks daily administration Cereal 2

INTERVENTIONS:
Dietary Supplement: 12 weeks daily administration Cereal 1 — The subjects will come to a visit every 4 weeks for a total period of 12 weeks. At the first, the second and the third visit the subjects will be supplied with a 5-week supply of product.
  Each daily administration will be supplied in a sachet. Subjects will be instructed to mix the contents of the sachet with 200mL of water and drink the solution within 5 minutes after preparation.
  The daily dose administrated is 15 grams.
  Arms: 12 weeks daily administration Cereal 1
Dietary Supplement: 12 weeks daily administration Cereal 2 — The subjects will come to a visit every 4 weeks for a total period of 12 weeks. At the first, the second and the third visit the subjects will be supplied with a 5-week supply of product.
  Each daily administration will be supplied in a sachet. Subjects will be instructed to mix the contents of the sachet with 200mL of water and drink the solution within 5 minutes after preparation.
  The daily dose administrated is 15 grams.
  Arms: 12 weeks daily administration Cereal 2
Other: 12 weeks daily administration Placebo — The subjects will come to a visit every 4 weeks for a total period of 12 weeks. At the first, the second and the third visit the subjects will be supplied with a 5-week supply of placebo.
  Each daily administration will be supplied in a sachet. Subjects will be instructed to mix the contents of the sachet with 200mL of water and drink the solution within 5 minutes after preparation.
  Arms: 12 weeks daily administration Placebo

SUMMARY:
This study evaluates the effect in HbA1c levels of a once daily administration of plant-based hydrolysates in pre-diabetic, but otherwise healthy volunteers. Among the 63 subjects enrolled, 21 will receive a plant-based hydrolysates from one cereal, 21 will receive a plant-based hydrolysates from another cereal and 21 will receive a placebo.

DETAILED DESCRIPTION:
Pre-clinical data on human skeletal muscle cells and mouse Type 2 diabetes model have shown a blood glucose lowering effect of the plant-based hydrolysates.

The first objective of the study is to evaluate the effect of a once daily administration of 2 different cereal protein hydrolysates versus placebo, when consumed over a 12-week period, at reducing the preferred outcome measure identified by the European Food Safety Authority i.e. glycated haemoglobin (HbA1c) levels in pre-diabetic volunteers who are otherwise healthy subjects.

The second objective of the study is to evaluate the effect of a fixed daily administration of 2 different cereal protein hydrolysates versus placebo, when consumed over a 12-week period on further supportive measures like Post-prandial glucose/insulin levels, fructosamine level, fasting plasma glucose level, vital signs and blood pressure, weight and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent,
* Be aged between 18 and 75 years, inclusive,
* Have a HbA1c of > 5.7% and < 6.4% (38.8mmol/mol- 47mmol/mol),
* Be a non-smoker or an ex-smoker (10 years or more),
* Have a body mass index (BMI) 20 - 35 kg/m²,
* Have a stable bodyweight (+/- 5%) in the last 3 months (as self-reported by the subject),
* Be willing to maintain existing dietary habits and physical activity levels throughout the trial period,
* Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator.

Exclusion Criteria:

* Diagnosed diabetes with a HbA1c >6.4% (47mmol/mol)
* Body Mass Index (BMI) less than 20 (underweight) or greater than 35 (morbidly obese)
* Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigators judgement, entry to the study
* Consumption of more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females
* Currently or recently (within 3 months of study entry) taking any medication, which in the opinion of the investigator, could interfere with the outcome of the study, including insulin, acetylsalicylic acid, thyroxine etc.
* If subjects are taking hypolipidemic agents and/or beta-blockers
* Known allergy to any of the components of the test product
* History of drug or alcohol abuse
* Present or recent use (within 3 months of pre-screening) of dietary supplements that may affect the level of blood glucose, e.g. chromium, dietary fibres and non-digestible carbohydrates e.g. fructo-oligosaccharides chicory inulin, mulberry leaf extract, e.t.c (Note: There are many dietary supplements, both approved and unapproved, marketed for the regulation of blood glucose. The Principal Investigator will discuss any uncertain cases directly with the study sponsor prior to inclusion of any such subjects)
* Low hemoglobin or hematocrit (i.e., lower than normal ranges specified and in-use at the local laboratory designated for this study),
* Females are pregnant, lactating or wish to become pregnant during the study.
* Participation in a clinical trial with an investigational product within 90 days before pre-screening, or plans to participate in another study during the study period,
* Subject has a history of non-compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Effect of the treatment on reduction of the HbA1c level (%) | 12 weeks
  Evaluate the effect of a once daily administration of the cereal 1 or cereal 2 protein hydrolysate versus placebo, when consumed over a 12-week period, at reducing the HbA1c level (%).

SECONDARY OUTCOMES:
Effect of the treatment on evolution of another parameter related to pre-diabetic condition: post-prandial glucose level | 12 weeks
  Evaluate the effect of a once daily administration of the cereal 1 or cereal 2 protein hydrolysate versus placebo, when consumed over a 12-week period, at reducing the post-prandial glucose level (mmol/L).
Effect of the treatment on evolution of another parameter related to pre-diabetic condition: post-prandial insulin level | 12 weeks
  Evaluate the effect of a once daily administration of the cereal 1 or cereal 2 protein hydrolysate versus placebo, when consumed over a 12-week period, at modifying the post-prandial insulin level (microU/mL).
Effect of the treatment on evolution of another parameter related to pre-diabetic condition: fructosamine level | 12 weeks
  Evaluate the effect of a once daily administration of the cereal 1 or cereal 2 protein hydrolysate versus placebo, when consumed over a 12-week period, at modifying the fructosamine level (microU/mL).
Effect of the treatment on evolution of the subject weight | 12 weeks
  Evaluate the effect of a once daily administration of the cereal 1 or cereal 2 protein hydrolysate versus placebo, when consumed over a 12-week period, at reducing the weight (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Valdis Pirags, Prof., Principal Investigator — P. Stradins University Hospital
Locations (2):
- Latvia (2):
  - P. Stradins Clinical University Hospital, Riga, LV
  - Clinic "Adoria" SIA, Riga, LV

IPD SHARING:
Plan to Share IPD: Undecided